CLINICAL TRIAL: NCT02191267
Title: Tau Imaging of Chronic Traumatic Encephalopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); Boston University (Other)
Responsible Party: Principal Investigator, Martha E Shenton, Director, Psychiatry Neuroimaging Laboratory, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014P000035
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-04

CONDITIONS: Chronic Traumatic Encephalopathy
Keywords: CTE; Positron Emission Topography; Tau; Beta-amyloid; Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy; Diffusion Tensor Imaging
MeSH Terms: conditions — Chronic Traumatic Encephalopathy; Pick Disease of the Brain; Plaque, Amyloid | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole; florbetapir; Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy; Diffusion Tensor Imaging; Genetic Testing; tau Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Presumed CTE Group (Experimental): Interventions administered to the Presumed CTE Group include: [F-18]-T807 PET Scan, [F18]-Florbetapir PET Scan, MRI/MRS Scans, and Genetic Analysis for Genetic Risk Score for Tau.
  Interventions: Radiation: [F18]-T807; Radiation: [F18]-Florbetapir; Device: MRI/MRS; Genetic: Genetic Analysis for Genetic Risk Score for Tau.
- Control Group (Experimental): Interventions administered to the Control Group include: [F-18]-T807 PET Scan, [F18]-Florbetapir PET Scan, and MRI/MRS Scans.
  Interventions: Radiation: [F18]-T807; Radiation: [F18]-Florbetapir; Device: MRI/MRS
- AD Dementia Group (Experimental): Interventions administered to the AD Dementia Group include: [F-18]-T807 PET Scan, [F18]-Florbetapir PET Scan, MRI/MRS Scans
  Interventions: Radiation: [F18]-T807; Radiation: [F18]-Florbetapir; Device: MRI/MRS

INTERVENTIONS:
Radiation: [F18]-T807 — [F18]-T807 PET Scan to measure tau deposition in the brain.
  Other Names: [F-18] AV-1451
Radiation: [F18]-Florbetapir — [F18]-Florbetapir PET scan to measure Beta-amyloid deposition in the brain.
  Other Names: Amyvid
Device: MRI/MRS — Two scans (structural, diffusion tensor imaging, and susceptibility weighted imaging scanned as part of one MR protocol, and a one-dimensional and two-dimensional spectroscopy examination as part of the other MR protocol.
  Other Names: Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy; Diffusion Tensor Imaging; Susceptibility Weighted Imgaging; One-dimensional Spectroscopy; Two-dimensional Spectroscopy
Genetic: Genetic Analysis for Genetic Risk Score for Tau. — DNA will be extracted from previously acquired and de-identified frozen blood specimens using a standard protocol (Gentra Puregene Kit, Qiagen 158422). Genotyping will be performed using the iPLEX Sequenom MassARRAY platform and samples will be genotyped for single nucleotide polymorphisms (SNPs) associated with the deposition of neurofibrillary tangles.
  Arms: Presumed CTE Group

SUMMARY:
Chronic traumatic encephalopathy (CTE) is a progressive degenerative brain disease with symptoms that include memory loss, problems with impulse control, and depression that can lead to suicide. As the disease progresses, it can lead to dementia. Currently CTE can only be diagnosed postmortem where an over-accumulation of a protein called tau is observed. There is now a new experimental measure that makes it possible, for the first time, to measure tau protein in the living human brain using a novel positron emission tomography (PET) ligand, [F-18] AV-1451 (aka, [18F]-T807).

The main objective of this study is to use a novel PET approach to measure tau accumulation in the brain. The presence of CTE at autopsy in deceased National Football League (NFL) players has been well documented. Accordingly, we will conduct this study in a group of retired NFL players who have clinical symptoms of CTE and are suspected of having CTE based on high levels of tau in their spinal fluid and abnormalities seen on research brain scans. We will compare them with a control group of former elite level athletes who have not experienced any brain trauma, deny any clinical symptoms, and who have completely normal spinal fluid tau and amyloid levels, and brain scans. We will also include a group of subjects with AD. All participants will be recruited from ongoing studies, headed by the Partnering PI of this proposal, Dr. Robert Stern, at the Boston University Center for the Study of Traumatic Encephalopathy and the Alzheimer's Disease Center. We will use both a beta amyloid PET scan ([18F]-florbetapir) and a tau PET scan ([18F]-T807) on consecutive days. With the beta amyloid scan we expect little or no evidence of amyloid in the NFL players with presumed CTE, and no evidence of amyloid in the control group of athletes with no history of repetitive brain trauma. In contrast we expect to see beta amyloid accumulation in the AD patient brains. With the new tau ligand, we expect that the NFL players with presumed CTE will show elevated levels of tau protein in the brain, which will not be observed in athletes without a history of brain trauma, but which will be seen in the AD patients' brains.

Another goal is to use the latest MRI technologies to develop specific tau imaging biomarkers that correlate with the PET and spinal fluid tau measures but without the radiation of PET or invasiveness of spinal taps. The development of these surrogate imaging markers of tau, is critically important to diagnosing CTE. This in turn will lead to studies relevant to treatment and prevention of this devastating disease. Finally, as an exploratory method of examining possible genetic risk for CTE, we will also use cutting edge genetic analysis of blood samples from subjects in this proposal and compare tau load, measured by PET tau ligand uptake and cerebrospinal fluid (CSF) p-tau level, with a measure of genetic susceptibility to tau load, referred to as the genetic risk score for tau.

ELIGIBILITY:
1. Presumed CTE Group (includes 20 former NFL players who will have already participated in the NIH-funded R01 "DETECT" (Diagnosis and Evaluation of Traumatic Encephalopathy with Clinical Tests) study (Stern, PI; Shenton, Neuroimaging Site PI). Eligibility criteria for presumed CTE group and the control group are based on findings from the DETECT study.

   Inclusion Criteria:
   * significant cognitive impairment (and impairment in at least one of the following):
   * behavioral (e.g., impulsivity, aggression),
   * mood (e.g., elevated depression measures, elevated suicidality),
   * and/or motor (e.g., impairments evidenced in neurological examination;
   * demonstrated abnormalities on svMRI, DTI, or MRS

   Exclusion Criteria:
   * weight > 350 lbs
   * known metallic implants preventing MRI
   * history of stroke
   * non-English speaking
   * significant vision or hearing impairment
   * unable to provide written informed consent
2. Control Group (comprised of 5 male participants selected from 50 control subjects in the DETECT study).

   Inclusion Criteria:
   * no history of mTBI or exposure to repetitive brain trauma
   * normal functioning on DETECT clinical measures
   * no abnormalities on svMRI, DTI, or MRS

   Exclusion Criteria:
   * weight > 350 lbs
   * known metallic implants preventing MRI
   * history of stroke or other neurological disease
   * non-English speaking
   * significant vision or hearing impairment
3. AD Dementia Group (comprised of 5 male participants recruited from the BU Alzheimer's Disease Center (ADC) Clinical Core Registry (Dr. Stern, PI).

Inclusion Criteria:

* diagnosis of Dementia due to AD using the NIA-AA (National Institute on Aging-Alzheimer's Association) criteria
* Clinical Dementia Rating Global Score of 1.0,
* a positive florbetapir PET study,
* CSF p-tau/Aβ consistent with AD.

Exclusion Criteria:

* history of TBI, mTBI or or exposure to repetitive brain trauma
* weight > 350 lbs
* known metallic implants preventing MRI
* history of stroke or other neurological disease
* non-English speaking
* significant vision or hearing impairment

Ages: 40 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha E. Shenton, Ph.D., Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Boston University Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

REFERENCES:
- [Background] Zhang W, Arteaga J, Cashion DK, Chen G, Gangadharmath U, Gomez LF, Kasi D, Lam C, Liang Q, Liu C, Mocharla VP, Mu F, Sinha A, Szardenings AK, Wang E, Walsh JC, Xia C, Yu C, Zhao T, Kolb HC. A highly selective and specific PET tracer for imaging of tau pathologies. J Alzheimers Dis. 2012;31(3):601-12. doi: 10.3233/JAD-2012-120712. PMID 22683529
- [Background] Chien DT, Bahri S, Szardenings AK, Walsh JC, Mu F, Su MY, Shankle WR, Elizarov A, Kolb HC. Early clinical PET imaging results with the novel PHF-tau radioligand [F-18]-T807. J Alzheimers Dis. 2013;34(2):457-68. doi: 10.3233/JAD-122059. PMID 23234879

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 subjects at presumed risk for Chronic Traumatic Encephalopathy (CTE), 6 healthy control subjects without a history of repetitive brain trauma, and 4 Alzheimer's Disease (AD) subjects were recruited from the Boston University Center for the study of Chronic Traumatic Encephalopathy.
Pre-assignment Details: Subjects were pre-assigned according to previously assigned study diagnostic status based on prior participation in studies at the Boston Center for the study of Chronic Traumatic Encephalopathy.
Groups:
- Presumed CTE Group: Interventions administered to the Presumed CTE Group include: [F-18]-T807 PET Scan and [F18]-Florbetapir PET Scan.
  [F18]-T807: [F18]-T807 PET Scan to measure tau deposition in the brain.
  [F18]-Florbetapir: [F18]-Florbetapir PET scan to measure Beta-amyloid deposition in the brain.
- Control Group: Interventions administered to the Control Group include: [F-18]-T807 PET Scan and [F18]-Florbetapir PET Scan.
  [F18]-T807: [F18]-T807 PET Scan to measure tau deposition in the brain.
  [F18]-Florbetapir: [F18]-Florbetapir PET scan to measure Beta-amyloid deposition in the brain.
- AD Dementia Group: Interventions administered to the AD Dementia Group include: [F-18]-T807 PET Scan and [F18]-Florbetapir PET Scan.
  [F18]-T807: [F18]-T807 PET Scan to measure tau deposition in the brain.
  [F18]-Florbetapir: [F18]-Florbetapir PET scan to measure Beta-amyloid deposition in the brain.
Period: Overall Study
Arm/Group | Presumed CTE Group | Control Group | AD Dementia Group
Started | 20 | 6 | 4
Completed | 19 | 6 | 4
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Presumed CTE Group | Control Group | AD Dementia Group | Total
Number analyzed (Participants) | 19 | 6 | 4 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 6 | 4 | 29
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 19 | 6 | 4 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 1 | 0 | 7
  White | 13 | 5 | 4 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 6 | 4 | 29

OUTCOME MEASURES:

1. Primary Outcome: Tau Protein Uptake..
Description: Whole brain mean (and standard deviation) cortical value derived from standardized uptake value ratio (SUVr). Each [F18]-T807 tau scan consisted of a 60-minute dynamic acquisition after bolus intravenous injection of 10 mCi of [18F]-T807, followed by a second 20-minute dynamic imaging (list mode) acquisition from 80-100 minutes. SUVr images were constructed from the sum of the 80-100 minute frames resulting in late SUVr distribution maps.
Time Frame: Day 1 - of 2 day study.
Measure: Mean (Standard Deviation); unit: SUVr
Arm/Group | Presumed CTE Group | Control Group | AD Dementia Group
Number analyzed (Participants) | 19 | 6 | 4
SUVr | 1.1871 (0.0762) | 1.1652 (0.0670) | 1.5910 (0.3807)

2. Secondary Outcome: Beta-Amyloid (Aβ) Protein Uptake.
Description: Mean and standard deviation for standardized uptake value ratios (SUVr) for posterior cingulate, superior parietal, lateral frontal, medial frontal, lateral temporal, and occipital brain regions. Each [F18]-Florbetapir (Beta-Amyloid) scan consisted of a 70-minute dynamic acquisition after bolus intravenous injection of 10 mCi of [18F]-Florbetapir. SUVr images were constructed from the sum of the 50-70 minute frames resulting in late SUVr distribution maps.
Time Frame: Day 2 - of 2 day study.
Measure: Mean (Standard Deviation); unit: SUVr
Arm/Group | Presumed CTE Group | Control Group | AD Dementia Group
Number analyzed (Participants) | 19 | 6 | 4
SUVr
  Posterior Cingulate | 1.346 (0.215) | 1.290 (0.068) | 1.760 (0.352)
  Superior Parietal | 1.225 (0.180) | 1.118 (0.073) | 1.708 (1.708)
  Lateral Frontal | 1.196 (0.178) | 1.145 (0.085) | 1.728 (0.291)
  Medial Frontal | 1.253 (0.190) | 1.182 (0.083) | 1.847 (0.261)
  Lateral Temporal | 1.178 (0.164) | 1.113 (0.083) | 1.766 (0.345)
  Occipital | 1.288 (0.191) | 1.157 (0.039) | 1.540 (1.540)

ADVERSE EVENTS:
Time Frame: Through study completion, Subjects were assessed for adverse effects immediately following each scan (On Day 1 and Day 2) and again by telephone 72 hours following study participation. Thus, assessment for adverse events were made over over a 5-day period which included Days 1 and 2 of the study visit and a follow-up telephone assessment on Day 5.
Arm/Group | Presumed CTE Group | Control Group | AD Dementia Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 0/19 | 0/6 | 0/4

LIMITATIONS AND CAVEATS:
Exploratory aims including potential MRI and MRS biomarkers and genetic analysis for genetic risk score for Tau will also be analyzed but are not primary or secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No